CLINICAL TRIAL: NCT01422278
Title: Patients With Conversion Gait Disorder - Effect on Treatment and Common Gait Patterns. Randomized Clinical Trial
Brief Title: Rehabilitation of Conversion Gait Disorder
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Annika A. Jordbru, PhD student, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2.2004.164; SSR.2005.1
Record Dates: First submitted 2006-01-16; First posted 2011-08-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Conversion Disorder
MeSH Terms: conditions — Conversion Disorder | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Rehabilitation — Three weeks of rehabilitation in Hospital.

SUMMARY:
Evaluating the effects in functional status after three weeks of cognitive - and behavioural rehabilitation on patients with gait disorder. The patients are followed up as after 1 and 12 months to study if any improvement is still present. The patients are being recruited from neurological units. The intervention is explanation of symptoms, positive reinforcement of normal behaviour and absence reinforcement of dysfunctional behaviour. In addition the study aims at describing typical gait patterns at patients with gait disorder by using biomechanical measurements (EKG).

DETAILED DESCRIPTION:
Patients are being recruited from neurological unit/ div and out patients department of SSR and are randomized to treatment or control group. Essential gait disorders do to conversion symptoms and willingness to participate in either of the two groups with informed consent are required.

ELIGIBILITY:
Inclusion Criteria:

* To determine the changes in functional status after three weeks of multidisciplinary rehabilitation in patients with conversion walking disorder.

Exclusion Criteria:

* Essential gait disorders do to conversion symptoms and willingness to participate in either of the two groups with informed consent are required.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change in gait patterns | three weeks

SECONDARY OUTCOMES:
Improved life quality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Høyer, DH, Study Chair — National committees for research ethics in Norway" for REK
Locations (1):
- Vestfold Hospital Trust, clinic physical medicine and rehabilitation, Stavern, Vestfold, Norway